CLINICAL TRIAL: NCT04133246
Title: Expectations and Needs of Patients With Cystic Fibrosis Becoming Parents - Exploratory Study
Brief Title: Parenting Concerns in Patients With Cystic Fibrosis (MucoPar)
Acronym: MucoPar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-A03241-54
Record Dates: First submitted 2019-09-04; First posted 2019-10-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; parenthood; Psycho-social; Qualitative study
MeSH Terms: conditions — Cystic Fibrosis | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group arm (Other): Includes subjects enrolled in focus groups
  Interventions: Behavioral: Focus group
- Interview arm (Other): Includes subjects with individual interviews
  Interventions: Behavioral: Individual interview

INTERVENTIONS:
Behavioral: Focus group — Groups of 6 to 10 patients and spouses led by the psychologist about their parenthood lasting 2 hours
  Arms: Group arm
Behavioral: Individual interview — Interview led by the psychologist about the patient's parenthood
  Arms: Interview arm

SUMMARY:
The purpose of this study is to explore and collect the perceptions, expectations and needs of CF patients about parenting. This will be done in the context of several small groups of patients led by a psychologist who will ensure that all the participants express themselves; he will encourage them to develop their points of view, their divergences and their common points about what constitutes to be a parent.

The collected information should make it possible to develop and propose adapted medico-psycho-social interventions, if necessary, in connection with patient associations

DETAILED DESCRIPTION:
Life expectancy has improved significantly in cystic fibrosis in recent years. From paediatric disease, it has become a disease of the adult, with the emergence of new issues, such as becoming a parent. Parent patients still face the risk of complications and death while their child is still young. However, there is very little data in the literature on parenting in cystic fibrosis.

Therefore, the purpose of this study is to explore and collect the perceptions, expectations and needs of CF patients and their spouses about parenting.

All patients with children, followed in 2 large adult CF centers, and their spouses will be invited to participate in a 6 to 10-person discussion group (focus group) led by a psychologist. He will ensure that all the participants express themselves and are encouraged to develop their points of view, their divergences and their common points about what constitutes to be a parent. The discussions will be recorded and transcribed.

Patients who cannot participate in groups (e.g. patients colonized with Burkholderia cepacia complex) but wish to be included in the study will benefit from an individual interview with the psychologist, also registered and transcribed. A thematic analysis will be carried out from the transcriptions of group contents. For individual interviews, phenomenological interpretative analysis (IPA) will be used. A synthesis of the two analyses will then be done.

The collected information should make it possible to develop and propose adapted medico-psycho-social interventions, if necessary, in connection with patient associations.

ELIGIBILITY:
Inclusion Criteria:

For patients

* Have cystic fibrosis
* Be a parent and raise or have raised at least one child
* Being followed in one of the two adult CF centers participating in the study

For CF patients' spouses

- Live with the CF patient participating in the study

For both CF patients and spouses

* Being an adult (at least 18 y.o.)
* Have a good level of French and good speaking skills

Exclusion Criteria:

* For both CF patients and spouses
* Psychiatric pathology (borderline state, bipolarity and other psychotic disorders)
* Serious somatic disease not related to cystic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Identification of themes about parenthood in CF from groups | 2 years
  by thematic analysis. 8 to 10 focus groups composed of 5 to 10 persons are to be conducted until saturation of themes.

SECONDARY OUTCOMES:
Identification of themes about parenthood in CF from individual interviews | 2 years
  by the IPA method. 20 individual interviews are to be conducted until saturation of themes
Occurrence of themes | 2 years
  number of appearances of each theme, revealed by the 2 analyses, in the group arm on one hand, and in the interview arm on the other hand. The occurrence will provide information on the importance of each theme

CONTACTS AND LOCATIONS:
Overall Officials: Cécile FLAHAULT, Ph.D, Study Chair — Assistance Publique - Hôpitaux de Paris; Dominique HUBERT, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Cochin Hospital, Paris, Île-de-France Region
  - Foch Hospital, Suresnes, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jacob A, Hubert D, Brain C, Grenet D, Flahault C. Exploring the lived experiences of parents living with cystic fibrosis: A qualitative study. J Health Psychol. 2025 Aug;30(9):2183-2200. doi: 10.1177/13591053241307874. Epub 2025 Jan 7. PMID 39764735